CLINICAL TRIAL: NCT07008573
Title: Prospective, Randomized, Multi-Center Comparative Study Evaluating the Efficacy of Topical Probiotics in Soyabean Concentrate in the Management of Diabetic Foot Ulcers
Brief Title: Prospective, Randomized, Multi-Center Comparative Study on Topical Probiotics in Diabetic Foot Ulcers
Status: Completed | Type: Observational
Sponsor: Tzu Chi University (Other)
Collaborators: Hualien Tzu Chi General Hospital (Other); Taichung Tzu Chi Hospital (Other)
Responsible Party: Principal Investigator, Honda Hsu, Associate Professor, Tzu Chi University
Other Study IDs: A11002001
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Diabetic Foot Ulcer
Keywords: probiotics; soybean concentrate
MeSH Terms: conditions — Diabetic Foot | interventions — Probiotics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment group: Treated with probiotics in soybean concentrate
  Interventions: Other: probiotics in soybean concentrate
- control group: Treated with placebo
  Interventions: Other: probiotics in soybean concentrate

INTERVENTIONS:
Other: probiotics in soybean concentrate — treatment with topical probiotics on DFU
  Other Names: Lactera

SUMMARY:
Looking at the efficacy of using Probiotics in Soyabean Concentrate in the management of diabetic lower extremity ulcers when administered by a wider variety of clinicians at multiple locations with a more heterogeneous patient

DETAILED DESCRIPTION:
Diabetic foot ulcers and pressure injury wounds are still a very common problem. According to International Diabetic Federation (IDF) around 12-15% of the general diabetic patient with develops a diabetic foot ulcer. These ulcers if not properly treated and managed can lead to major limb amputation. The 5-year survival rate according to our own previous study is around 67%. The management of the diabetic foot ulcer is at present being met using advanced wound care and surgical debridement and reconstruction.

Probiotics has recently being discussed as an effective form of management for these chronic wounds. Probiotics exert their positive effects through multiple mechanisms including: (a) competition with pathogenic bacteria for nutrients and binding sites on the host cell; (b) inactivation of toxins and metabolites, (c) production of antimicrobial substances that inhibit the growth of pathogenic microorganisms, and (d) stimulation/modulation of host immune response. Probiotic-host interactions involving epithelial cells (EC), dendritic cells (DC), and regulatory T lymphocytes have also been well studied particularly in the GI tract.

This study looks at the efficacy of using Probiotics in Soyabean Concentrate in the management of diabetic lower extremity ulcers when administered by a wider variety of clinicians at multiple locations with a more heterogeneous patient

ELIGIBILITY:
Inclusion Criteria:

* Age 20 or older Type 1 or Type 2 diabetes Able and willing to provide consent and agrees to comply with study procedures and follow-up evaluations Ulcer size 1cm2 and < 25cm2 Ulcer duration of 4 weeks, unresponsive to standard wound care Serum creatinine <3.0 mg/dL HBA1C <12% No clinical peripheral arterial occlusive disease. Able to carry out the wound care as described in the study

Exclusion Criteria:

* Current participation in another clinical trial Ulcer with exposure of tendon or bone Severely infected wound Currently under radio or chemotherapy Known or suspected malignancy of current ulcer Use of biomedical/topical growth factor within previous 30 days Pregnant or breast feeding Taking medications considered to be immune system modulators Allergy to known sensitivity to Probiotics of Soyabean. Inability to carry out wound care as described in the study. Inability to sign an informed consent form

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with diabetic foot ulcers without bone or tendon exposure with ulcer size between 1 cm² and < 25 cm²
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
incidence of complete wound closure at 24weeks. | 24 weeks

SECONDARY OUTCOMES:
time to healing and incidence of ulcer recurrence at the site of the study ulcer during the follow-up phase | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Honda Hsu, MBChB, Principal Investigator — Tzu Chi University
Locations (1):
- Dalin Tzu Chi Hospital, Dalin, Chaiyi, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT07008573/Prot_SAP_000.pdf